CLINICAL TRIAL: NCT00219531
Title: Effect of Menstrual Cycle and Irritable Bowel Syndrome on the Central Nervous System Processing of Gut Stimuli
Brief Title: Effect of Menstrual Cycle on Central Nervous System (CNS) Processing of Gut Stimuli in Irritable Bowel Syndrome (IBS) and Control
Status: Terminated | Type: Observational
Why Stopped: inadequate number of patients, study completed with normal subjects
Sponsor: Penn State University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); American College of Gastroenterology (Other)
Responsible Party: Sponsor
Other Study IDs: 99-073; NIDDK R21 DK57053; ACG Research Award 2000-2001
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Irritable Bowel Syndrome
Keywords: functional MRI; pain perception; anxiety; brain-gut axis
MeSH Terms: conditions — Irritable Bowel Syndrome; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- control: subjects with no irritable bowel syndrome or gastrointestinal complaints and regular menstrual cycle.
  Interventions: Behavioral: perception of rectal balloon distention
- IBS: women with IBS symptoms and normal menstrual cycle.
  Interventions: Behavioral: perception of rectal balloon distention

INTERVENTIONS:
Behavioral: perception of rectal balloon distention — functional Magnetic Resonance Imaging (fMRI) study with measurement of brain MRI response to rectal balloon distention.

SUMMARY:
The hypothesis of the study is that women perceive intestinal stimulation (rectal balloon distention) differently in different phases of the menstrual cycle, i.e there is an effect of hormones on the sensory pathway, and that this difference is reflected in the Central Nervous System processing of this signal. We also hypothesize that there is a difference in perception between control subjects and subjects with the irritable bowel syndrome.

DETAILED DESCRIPTION:
There is discrepancy in the literature concerning the effect of the menstrual cycle on bowel function and pain syndromes such at irritable bowel syndrome. In addition, recent studies indicate a difference in the CNS processing of rectal stimulation in normal subjects and patients with IBS. This study will determine the differences in the perception of rectal balloon distention in the follicular and luteal phases of the menstrual cycle, in control subjects with no bowel symptoms and volunteers with IBS, and will compare the CNS processing of this signal using functional MRI , again in the two phases of the menstrual cycle.

Comparisons: between control subjects without GI symptoms and those with irritable bowel syndrome.

ELIGIBILITY:
Inclusion Criteria:

* controls - normal bowel function
* Irritable bowel syndrome - Rome II criteria
* Normal menstrual cycle

Exclusion Criteria:

* irregular menses
* pregnancy
* use of psychotropic medication
* claustrophobia
* metal implants
* metal in eyes

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women with menstrual cycle
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 1999-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Sensitivity to rectal distention | during the study period only
  pressure at which certain sensations are felt when barostat is inflated in the rectum during follicular and luteal phase of menstrual cycle

CONTACTS AND LOCATIONS:
Overall Officials: Ann Ouyang, MD, Principal Investigator — Penn State College of Medicine and Penn State Milton S. Hershey Medical Center
Locations (1):
- Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Wrzos HF, Li Q, Ouyang A. Visceral and somatic pain thresholds in healthy and IBS volunteers across the menstrual cycle. The American Journal of Gastroenterology 98: S265, 2003